CLINICAL TRIAL: NCT04777760
Title: Surfactant for Neonatal Respiratory Distress Syndrome(NRDS) and Neonatal Acute Respiratory Distress Syndrome(NARDS)
Status: Recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, director, Children's Hospital of Chongqing Medical University
Other Study IDs: surfactant for NRDS and ARDS
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Distress Syndrome; Preterm Birth; Acute Respiratory Distress Syndrome; Surfactant Dysfunction
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth; Surfactant Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- one dose of surfactant: the preterm infants diagnosed with NRDS and/or NARDS will be administrated with only one dose of surfactant
  Interventions: Drug: one dose of surfactant replacement
- two and more doses of surfactant: the preterm infants diagnosed with NRDS and/or NARDS will be administrated with two and more doses of surfactant
  Interventions: Drug: two and more doses of surfactant replacement

INTERVENTIONS:
Drug: one dose of surfactant replacement — the preterm infants diagnosed with NRDS and/or NARDS will be administrated with only one dose of surfactant
  Groups: one dose of surfactant
Drug: two and more doses of surfactant replacement — the preterm infants diagnosed with NRDS and/or NARDS will be administrated with two and more doses of surfactant
  Groups: two and more doses of surfactant

SUMMARY:
In preterm infants with neonatal respiratory distress syndrome (NRDS), exogenous pulmonary surfactant(PS) replacement therapy is one of the most important therapeutic breakthrough to reduce neonatal mortality. Nowadays, PS is commonly used in newborn infants with respiratory distress, but the incidences of bronchopulmonary dysplasia(BPD) and/or death are inconsistent. The result indicates that not all preterm infants with respiratory distress can be beneficial from PS.

In 2017, the international neonatal ARDS (NARDS) collaborative group provides the first consensus definition for NARDS. And whether or not PS being beneficial for preterm infants with NARDS remains unknown.

DETAILED DESCRIPTION:
To date, PS is not recommended to adult and pediatric ARDS. Meantime, systematic review indicates that PS does not demonstrate statistically significant beneficial effects on reducing the mortality and the rate of BPD in term and late preterm infants with meconium aspiration syndrome(MAS). Therefore, a reasonable speculation is that preterm infants with NARDS do not benefit from one dose of PS. And the speculation can explain why not all preterm infants with respiratory distress can be beneficial from PS. In the era of pre-NARDS, the preterm infants fulfilling the definition of NARDS may have been considered as NRDS in the first three days after birth.

According to the diagnostic criteria of NARDS, a key procedure for diagnosis of NARDS is to exclude the newborn infants with NRDS. But no detailed procedures are available to differentiate NRDS from NARDS.

ELIGIBILITY:
Inclusion Criteria:

Eligibility requirements for neonates were as follows:

* The gestational age is less than 37 weeks and admitted to neonatal intensive care unit(NICU) in 24 h after birth
* The neonates will be diagnosed with NRDS or NARDS
* The neonates will be at least administrated one dose of surfactant

Exclusion Criteria:

one of the following criteria will be needed

* major congenital anomalies
* chromosomal abnormalities
* upper respiratory tract abnormalities

Ages: 1 Minute to 24 Hours | Sex: All
Age Groups: Child
Study Population: Preterm infants diagnosed with NRDS or NARDS were eligible. The diagnosis of NARDS was according to the criteria established by Montreux conference in 2017.The diagnosis of NRDS was according to the criteria established by European Consensus Guideline for the management of NRDS in 2019
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
bronchopulmonary dysplasia(BPD) | at 36 weeks' gestational age or before discharge from hospital
  the preterm infants will be diagnosed with BPD
death | at 36 weeks' gestational age or before discharge from hospital
  the preterm infants die
BPD and/or death | at 36 weeks' gestational age or before discharge from hospital
  the preterm infants will be diagnosed with BPD and/or death
the predictive powers of one dose of surfactant to diagnose NRDS | seven days after birth
  the sensitivity and accuracy of one dose of surfactant to diagnose NRDS
the predictive powers of two and more doses of surfactant to diagnose NARDS | seven days after birth
  the sensitivity and accuracy of two and more doses of surfactant to diagnose NARDS

SECONDARY OUTCOMES:
intraventricular hemorrhage(IVH) | before discharge or 36 weeks' gestational age
  the preterm infants will be diagnosed with IVH
air leak | at 36 weeks' gestational age or before discharge from hospital
  the preterm infants will be diagnosed with air leak
periventricular leukomalacia(PVL) | at 36 weeks' gestational age or before discharge from hospital
  the preterm infants will be diagnosed with PVL
necrotizing enterocolitis(NEC) | at 36 weeks' gestational age or before discharge from hospital
  the preterm infants will be diagnosed with NEC
patent ductus arteriosis(PDA) | at 36 weeks' gestational age or before discharge from hospital
  the preterm infants will be diagnosed with PDA
late-onset sepsis(LOS) | at 36 weeks' gestational age or before discharge from hospital
  the preterm infants will be diagnosed with LOS

CONTACTS AND LOCATIONS:
Locations (1):
- Chen, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
the data will be accessed after two years of study accomplishment
Supporting Information: Study Protocol, SAP, CSR
Time Frame: preliminary estimate in 2025